CLINICAL TRIAL: NCT05921058
Title: The Effects of Mesenchymal Stem Cell Secretome in Lupus Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Arief Nurudhin, MD. Ph.D, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAP05
Record Dates: First submitted 2023-03-09; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Lupus Erythematosus
Keywords: Messenchymal Stem Cell Secretome; Lupus
MeSH Terms: interventions — Secretome

STUDY DESIGN:
Intervention Model Description: This study was divided into two groups, namely, control and treatment. Both received intervention in the form of a 1.5 cc injection on the scheduled day
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Mesenchymal stem cell placebo and secretome using injections that are similar in shape and color
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Messenchymal stem cell secretome (Experimental): The hypoxic mesenchymal stem cell secretome has been developed up to chapter 7, stored at -196 C to -135 C in cryopreservation, and has passed quality tests.
  Interventions: Drug: Secretome
- Placebo (Placebo Comparator): Nacl 0,9% infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secretome — Mesenchymal stem cell secretome obtained from Kalbe Pharma Company
  Other Names: Messenchymal stem cell Concitioned Media
  Arms: Messenchymal stem cell secretome
Drug: Placebo — NaCl 0,9% infusion
  Other Names: NaCl 0,9% infusion
  Arms: Placebo

SUMMARY:
This research is a clinical trial of administering mesenchymal stem cell secretome to lupus patients.

DETAILED DESCRIPTION:
This research is experimental. The study was conducted on 30 SLE patient subjects. the treatment group who got the mesenchymal stem cell secretome on the 1st, 2nd day, 3rd, 4th, 5th, 6th, 7th, 14th, 21st, and 28th days. ESR, hs-CRP, C3, C4, interlukin 6, anti-ds-DNA antibody, MEX SLEDAI score, and assessment of drug side effects before and after therapy were collected. Statistical test with paired difference test with p < 0.05

ELIGIBILITY:
Inclusion Criteria:

* Lupus paatients

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Lupus Disease activity | Change of Lupus Disease Activity at 1 months
  The data collected were MEX SLEDAI score (range 0-32) before and after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nurhasan Agung Prabowo, MD, Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Moewardi General Hospital, Surakarta, Middle Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pratama YS, Pradiptakirana R, Rachmah A, Prabowo NA. Autoimmune Thrombocytopenia in SLE and COVID-19. Eur J Case Rep Intern Med. 2021 Nov 3;8(11):002863. doi: 10.12890/2021_002863. eCollection 2021. PMID 34912736
- [Result] Sholihah MM, Kusuma TRH, Hanif MI, Prabowo NA. Letter to the Editor on Type 1 diabetes onset triggered by COVID-19. Acta Diabetol. 2021 Sep;58(9):1283-1284. doi: 10.1007/s00592-021-01761-3. Epub 2021 Jun 28. No abstract available. PMID 34181079